CLINICAL TRIAL: NCT02401256
Title: Influence of Autoinhibition/Autoinduction and CYP2B6 Genetic Variations on CYP2B6 Activity and Drug Interactions in Healthy Volunteers
Brief Title: CYP2B6 Genetics and Drug Interactions in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Principal Investigator, Zeruesenay Desta, Research Professor, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1205008739; 5R01GM078501 (NIH)
Record Dates: First submitted 2015-02-26; First posted 2015-03-27 (Estimated); Results first posted 2017-10-11 (Actual); Last update posted 2017-10-11 (Actual); Status verified 2017-09

CONDITIONS: Healthy
Keywords: Efavirenz; metabolism; pharmacokinetics changes
MeSH Terms: interventions — efavirenz; Bupropion; Rosuvastatin Calcium; montelukast

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CYP2B6 (Experimental): This is a fixed-order, open label prospective cohort study to determine: a) the contribution of CYP2B6 autoinhibition/autoinduction processes to variable CYP2B6 activity and efavirenz exposure; b) the impact of CYP2B6 genetic variants on these processes; and c) drug interactions that ensue.
  Included drugs:
  Efavirenz (600mg) - The volunteers will receive it in two of three inpatient visits and also during 17 days at home
  Bupropion (100mg), Montelukast (10mg) and Rosuvastatin (5mg) - These drugs will be administrated on 3 occasions (at the begging each inpatient visit of Phase 1, 2 and 4).
  Interventions: Drug: Efavirenz; Drug: Bupropion; Drug: Rosuvastatin; Drug: Montelukast

INTERVENTIONS:
Drug: Efavirenz — The study has 4 phases:
  Phase 1 (control)-Subjects will receive simultaneously a single dose of bupropion 100 mg, montelukast 10 mg and rosuvastatin 5 mg (cocktail) by mouth (control).
  Phase 2 (inhibition)- a single 600 mg oral dose of efavirenz (blood draw at 30 min and 1 hour) will be administered with the cocktail drugs.
  Phase 3 (home treatment with efavirenz): Subjects will take efavirenz at home (600 mg/day for 17 days).
  Phase 4 (Induction) - is the same as phase 2. Blood samples (0 to 120 hrs) and urine voided over 48 hrs (Phases 1, 2 and 4) are collected. Blood draws will be made in phase 3 for trough concentration measurements.
  Other Names: Sustiva
Drug: Bupropion — The study has 4 phases:
  Phase 1 (control)-Subjects will receive simultaneously a single dose of bupropion 100 mg, montelukast 10 mg and rosuvastatin 5 mg (cocktail) by mouth (control).
  Phase 2 (inhibition)- a single 600 mg oral dose of efavirenz (blood draw at 30 min and 1 hour) will be administered with the cocktail drugs.
  Phase 3 (home treatment with efavirenz): Subjects will take efavirenz at home (600 mg/day for 17 days).
  Phase 4 (Induction) - is the same as phase 2. Blood samples (0 to 120 hrs) and urine voided over 48 hrs (Phases 1, 2 and 4) are collected. Blood draws will be made in phase 3 for trough concentration measurements.
  Other Names: Wellbutrin
Drug: Rosuvastatin — The study has 4 phases:
  Phase 1 (control)-Subjects will receive simultaneously a single dose of bupropion 100 mg, montelukast 10 mg and rosuvastatin 5 mg (cocktail) by mouth (control).
  Phase 2 (inhibition)- a single 600 mg oral dose of efavirenz (blood draw at 30 min and 1 hour) will be administered with the cocktail drugs.
  Phase 3 (home treatment with efavirenz): Subjects will take efavirenz at home (600 mg/day for 17 days).
  Phase 4 (Induction) - is the same as phase 2. Blood samples (0 to 120 hrs) and urine voided over 48 hrs (Phases 1, 2 and 4) are collected. Blood draws will be made in phase 3 for trough concentration measurements.
  Other Names: Crestor
Drug: Montelukast — The study has 4 phases:
  Phase 1 (control)-Subjects will receive simultaneously a single dose of bupropion 100 mg, montelukast 10 mg and rosuvastatin 5 mg (cocktail) by mouth (control).
  Phase 2 (inhibition)- a single 600 mg oral dose of efavirenz (blood draw at 30 min and 1 hour) will be administered with the cocktail drugs.
  Phase 3 (home treatment with efavirenz): Subjects will take efavirenz at home (600 mg/day for 17 days).
  Phase 4 (Induction) - is the same as phase 2. Blood samples (0 to 120 hrs) and urine voided over 48 hrs (Phases 1, 2 and 4) are collected. Blood draws will be made in phase 3 for trough concentration measurements.
  Other Names: Singulair

SUMMARY:
The CYP2B6 enzyme metabolizes a growing number of clinically important drugs such as the anti-HIV drug efavirenz, but its activity in the liver is highly variable, which may lead to failure of therapy or toxicity and unpredictable drug interactions. Genetic and several nongenetic factors affect the activity of CYP2B6. The goal of this study is to determine the impact of simultaneous autoinhibition/autoinduction and CYP2B6 genetics on CYP2B6 activity, efavirenz exposure and efavirenz-mediated drug interactions. The pharmacokinetics and drug interactions will be determined on three occasions in a total of 60 healthy volunteers. The whole study will have 4 phases. A) Phase 1 (baseline control): using selective probe substrates, the baseline activities of CYP2B6 (bupropion), CYP2C8 (montelukast) and OATP1B1 (rosuvastatin) are determined. B) Phase 2 (inhibition): the metabolism and pharmacokinetics of a single 600 mg oral dose of efavirenz) and the activities of CYP2B6, CYP2C8 and OATP1B1 (inhibition) are determined. C) Phase 3 (treatment phase): After completing phase 2, subjects take 600 mg/day efavirenz at home for 17 days. C) Phase 4 (induction and inhibition): At the end of phase 3, steady state metabolism and pharmacokinetics of efavirenz and the activities of CYP2B6, CYP2C8 and OATP1B1 will be determined. Efavirenz serves as a model substrate, inhibitor and inducer of CYP2B6 (and other drug disposition proteins). Bupropion 4-hydroxylation is an alternative in vivo probe of CYP2B6 activity and will be studied here in addition to the metabolism and pharmacokinetics of efavirenz.

DETAILED DESCRIPTION:
Schedule of assessment

PHASE 1 (CONTROL PHASE)

Phase 1 (day 1 to day 4): baseline (control) activities of CYP2B6, CYP2C8 and OATP1B1 will be measured using selective probe substrates. Eligible subjects will receive simultaneously a single 100 mg dose of bupropion (CYP2B6), a single 10 mg dose montelukast (CYP2C8) and a single 5 mg dose of rosuvastatin (OATP1B1) by mouth on empty stomach together at least 10 days before phase 2. Frequent plasma samples will be collected for 72 hours and urine for 48 hours after dosing. Safety assessment will be made for the first 24 hours. Phase 1 is completed after the last blood draw on day 4 (72 hours).

PHASE 2 (INHIBITION PHASE)

In phase 2 (days 11 to 16), the metabolism and pharmacokinetics of a single 600 mg oral dose efavirenz will be determined along with the activities of CYP2B6, CYP2C8 and OATP1B1. Subjects receive a single 600 mg oral dose of efavirenz and blood samples will be obtained at 30 min and 1 hour. Immediately after the 1 hour blood draw, the three probe drugs (10 mg montelukast, 100 mg bupropion, and 5 mg rosuvastatin) will be administered simultaneously. Frequent plasma samples will be collected for 120 hours and urine for 48 hours after efavirenz dosing. Safety assessment will be made for the first 24 hours. Phase 2 is completed after the last blood draw on day 16 (120 hours). Note: The additional time points (compared to phase 1) are needed because of the long elimination half-life of efavirenz.

PHASE 3 (EFAVIRENZ TREATMENT PHASE).

In phase 3 (days 16 to 32), subjects will take efavirenz (600 mg/day) every evening for 17 days (Note: Phase 3 starts when the subject takes the first dose that evening on Day 16). Prior to taking the evening dose, they will be requested to return to the Indiana Clinical Research Center on day 19, day 22, day 25, day 28 and day 31 for a brief outpatient visit to have vital signs checked, draw blood sample (~10 ml, approximately 2 teaspoonful), and to fill out the brief central nervous system (CNS) symptoms questionnaire. They will be reminded not to take the evening dose of efavirenz on these days until after their blood draw. Since efavirenz has a long half-life (~76 hours after single dose and ~50 at steady state), a total of 17 days of efavirenz treatment is required to achieve steady-state plasma concentrations of efavirenz and steady-state autoinduction of metabolism. Subjects will be instructed to take efavirenz at bed-time to minimize efavirenz-induced central nervous side effects. Minor rescheduling (±3 days) of the subject's fixed inpatient/outpatient visits will be allowed including adjusting the amount of study medication (up to 3 doses less or up to 3 doses more) to be given prior to the subject's 4th inpatient visit.

PHASE 4 (INHIBITION/INDUCTION PHASE)

In phase 4 (days 33 to 38), the steady-state metabolism and pharmacokinetics of efavirenz will be determined along the activities of CYP2B6, CYP2C8 and OATP1B1. The procedures described in phase 2 will be repeated. On day 38, an exit exam will be performed consisting of a repeat of a repeat of the screening laboratory tests including blood and urine tests. The study diary will be collected. Medication bottles with left over pills (if any) will be returned and pills remaining will be counted for compliance purposes. The total duration of the study will be 38 days.

ELIGIBILITY:
A total of 60 healthy female and male volunteers (18 to 49 years old) who meet all inclusion and exclusion criterion listed below will be enrolled to participate in this study. All subjects will sign an Institutional Review Board (IRB) approved written informed consent prior to participation in the study after subjects read and carefully explained of the study to them. Then, potential subjects will undergo a pre-enrollment screening examination (a maximum of six weeks prior to enrollment into the study) for any medical abnormalities which will include medical histories, vital signs and electrocardiography, demographic variables, and standard laboratory blood and urine tests. The screening will be performed at the Indiana Clinical Research Center. During the screening, a blood sample (15 ml) will be collected from each subject for laboratory tests and urine for urine analyses. An additional ∼10 ml will be obtained from each subject to extract genomic DNA for genotyping purposes.

INCLUSION CRITERIA:

* 18 to 49 years old healthy male and female participants within 32% of their ideal body weight
* Individuals who agree to refrain from taking any prescriptions medications, over-the-counter medications, hormonal agents, and herbal, dietary, and alternative supplements that may interact with the metabolism of those study drugs at least 2 weeks prior to the start of the study and until study completion
* Nonsmoker or individuals willing to refrain from smoking or use of tobacco or marijuana for at least one month prior to and until the completion of the study (the entire study lasts for approximately 38 days)

EXCLUSION CRITERIA:

* Are underweight (less than 114 lb) or overweight (BMI greater than 32)
* Have history or current alcohol or drug abuse (more than 4 alcoholic drinks per day on a regular basis)
* Have history of intolerance, allergic reactions (e.g. rash) or other forms of hypersensitivities to any of the study medications (efavirenz, montelukast, bupropion and rosuvastatin)
* Have history or current significant health conditions such as heart, liver, or kidney
* Have history or current psychiatric illness such as depression, anxiety, or nervousness that may be exacerbated by participation in study
* Have a history of suicidality including suicide attempts
* Have history or current gastrointestinal disorders such as persistent diarrhea or malabsorption that would interfere with the absorption of orally administered drugs
* Have a serious infection within the last week before study enrollment
* Have a baseline EKG readings that is abnormal that could place the patient at the higher risk as decided by the study medical doctor (MD)
* Have donated blood within the past two months
* Have blood results that do not fall in a healthy range
* Are taking on regular basis substances that may interfere with the metabolism of study medications by the body, including prescription medications, over-the-counter, herbal or dietary supplements, alternative medications, or hormonal agents
* Are female with a positive pregnancy urine test obtained just prior to each study
* Are female breastfeeding
* Are child-bearing potential unable or unwilling to either practice abstinence or use two non-hormonal forms of birth control up until the study completion, which will take a total of 38 days
* Have a life style that places subjects at a higher risk for contracting HIV (e.g. drug abuse, excessive alcohol drinking, and having multiple sexual partners)
* Have a history or current HIV infection
* Have participation in a research study or use of an investigational drug in the last one month
* Are employed or are student under supervision of any of the investigators of this study
* Cannot state a good understanding of this study including risks and requirements; are unable to follow the rules of this study
* Cannot commit the time requested for this study

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Actual)
Dates: Start 2013-07; Primary Completion 2016-05 (Actual); Study Completion 2016-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Zeruesenay Desta, PhD, Principal Investigator — +1 (317) 274-2823
Locations (1):
- Indiana University School of Medicine, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 70 volunteers were enrolled study, 53 completed the whole study and 17 subjects withdraw from the study (6 during Phase 1, 6 during Phase 2 and 5 during Phase 3).
  We did include on the data analysis 8 volunteers that withdraw from the study but had Efavirenz quantification information and CYP2B6 genotypes (Analysed volunteers = 61)
Groups:
- CYP2B6: A cocktail of bupropion (100mg), montelukast (10mg) and rosuvastatin (5mg). These drugs will be administrated on 3 occasions (at the begging each inpatient visit of Phase 1, 2 and 4). The study has 4 phases: Phase 1 (control, baseline)Subjects received simultaneously a cocktail of a single dose of bupropion 100 mg (CYP2b6), montelukast 10 mg (CYP2C8) and rosuvastatin 5 mg (OATP1B1/BCRP) by mouth and their metabolism and pharmacokinetics determined. Phase 2 (inhibition)a single 600 mg oral dose of efavirenz is administered with the cocktail drugs listed above and their metabolism and pharmacokinetics determined Phase 3 (home treatment with efavirenz): Subjects is taken take efavirenz for approximately 17 days Phase 4 (induction): as in phase 2. Blood samples (0 to 120 hrs) and urine voided over 48 hrs (Phases 1, 2 and 4) are collected in all phases. Blood draws is made in phase 3 for trough concentration measurements.
Period: Overall Study
Arm/Group | CYP2B6
Started | 70
Finished Phase 1 | 64
Finished Phase 2 | 58
Finished Phase 3 | 53
Analysed | 61 (Volunteers that completed at least until Phase 2 inpatient visit (Volunteers with Efavirenz PK data))
Completed | 53
Not Completed | 17
Not completed — Adverse Event | 5
Not completed — Withdrawal by Subject | 12

BASELINE CHARACTERISTICS:
Arm/Group | CYP2B6
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 25.5 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 39
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8
  Not Hispanic or Latino | 62
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 14
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 12
  White | 40
  More than one race | 4
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Efavirenz AUC0-inf (Single Dose) and AUC0-24(Multiple Dose)
Description: After the samples collection, blood from phase 2 and phase 4 were used to perform the quantification of Efavirenz in plasma. The composite of the efavirenz concentration (blood collection between 0 to 120 hrs) were used to calculate the area under the plasma concentration time curve (AUC0-inf for single dose and AUC0-24 for multiple dose) of efavirenz.
Time Frame: Single dose pharmacokinetics (PK) versus multiple doses (after 17 day pretreatment) PK (total 38 days for each subject)
Population: Just volunteers with Efavirenz quantification information (complete or partial) and CYP2B6 genotype were included in this data analysis (Total of 61)
Measure: Mean (Standard Deviation); unit: h*uM
Groups:
- CYP2B6*1/*1; CYP2B6*1/*6; CYP2B6*6/*6: A cocktail of bupropion (100mg), montelukast (10mg) and rosuvastatin (5mg).These drugs will be administrated on 3 occasions (at the begging each inpatient visit of Phase 1, 2 and 4).The study has 4 phases:Phase 1(control/baseline).Subjects received simultaneously a cocktail of a single dose of bupropion 100 mg(CYP2B6), montelukast 10 mg(CYP2C8) and rosuvastatin 5 mg(OATP1B1/BCRP) by mouth and their metabolism and pharmacokinetics determined.Phase 2(inhibition)a single 600 mg oral dose of efavirenz is administered with the cocktail drugs listed above and their metabolism and pharmacokinetics determined Phase 3(home treatment with efavirenz):Subjects take efavirenz for approximately 17 days Phase 4 (induction): as in phase 2.Blood samples (0 to 120 hrs) and urine voided over 48 hrs(Phases 1, 2 and 4) are collected in all phases.Blood draws is made in phase 3 for trough concentration measurements. Volunteers were genotyped and stratified according to CYP2B6*1/*1, *1/*6, and *6/*6 alleles
Arm/Group | CYP2B6*1/*1 | CYP2B6*1/*6 | CYP2B6*6/*6
Number analyzed (Participants) | 22 | 33 | 6
h*uM
  Efavirenz AUC0-inf (Single Dose) | 411.53 (144.00) | 620.36 (269.12) | 522.42 (31.40)
  Efavirenz AUC0-24 (Multiple Dose) | 183.97 (62.49) | 254.40 (65.59) | 321.86 (146.28)

ADVERSE EVENTS:
Arm/Group | CYP2B6
All-Cause Mortality (participants affected / at risk) | 0/70
Serious Adverse Events (participants affected / at risk) | 0/70
Other Adverse Events (participants affected / at risk) | 5/70
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYP2B6 (N=70)
Efavirenz side effects (General disorders) | 5 (5) — Most common efavirenz side effects observed in this study: dizziness, nausea, vivid dreams, lack of concentration, headache, itching and rash (data collected using questionnaire and patient interview)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No